CLINICAL TRIAL: NCT00480363
Title: QUIREDEX: A National, Open-Label, Multicenter, Randomized, Phase III Study of Revlimid (Lenalidomide) and Dexamethasone (ReDex) Treatment Versus Observation in Patients With Smoldering Multiple Myeloma With High Risk of Progression
Brief Title: QUIREDEX: Revlimid (Lenalidomide) and Dexamethasone (ReDex) Treatment Versus Observation in Patients With Smoldering Multiple Myeloma With High Risk of Progression
Acronym: QUIREDEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Pethema, Pethema
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-000649-36; QUIREDEX
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma
Keywords: Smoldering Multiple Myeloma; PETHEMA; Smoldering
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Maintenance; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lenalidomide + Dexamethasone for 9 cycles and maintenance
  Interventions: Procedure: Maintenance with lower doses of lenalidomide and dexamethasone
- 2 (No Intervention): Observation

INTERVENTIONS:
Procedure: Maintenance with lower doses of lenalidomide and dexamethasone — After 9 cycles of lenalidomide and dexamethasone, it follows with lower doses for maintenance
  Arms: 1

SUMMARY:
The primary objective is to evaluate when Revlimid and Dexamethasone treatment extend the time to progression to symptomatic MM in patients with smoldering MM. The second one is to evaluate the efficacy of the treatment in response rate terms. Otherwise this study wants to evaluate the safety and tolerability of the treatment

DETAILED DESCRIPTION:
A total of up to 120 patients diagnosed of smoldering Multiple Myeloma with high risk of progression to symptomatic MM will be included.

Patients will be stratified according its diagnosis date and randomized 1 to 1 to receive Revlimid and Dexamethasone (Group A) in 9 treatment cycles and maintenance with lower doses until progression or No treatment and observation until progression (Group B).

The patients will be evaluated at scheduled visits in up to three study periods: Pre-treatment, Treatment and Follow up.

The Pre-treatment includes Screening and baseline visits. After providing informed consent, patients will be evaluated for study eligibility and then Patients will be stratified and randomized (1:1) to Group A or Group B.

During Treatment Period patients will be evaluated once a month. Once the treatment period has finished a maintenance treatment with low doses of Revlimid and Dexamethasone will be carry out in Group A. During this period we will evaluate response, progression-free survival and global survival every two months.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to comply with the protocol requirements
* Must voluntary sign the informed consent before performance of any study-related procedure not part of normal medical care
* Age ≥ 18 years
* Patient recently diagnosed with smoldering Multiple Myeloma with high risk of progression to symptomatic Multiple Myeloma defined as follows:

  * Bone Marrow infiltration ≥ 10% CPs and M component Ig G ≥ 3 g/dl or Ig A ≥ 2 g/dl or Bence Jones Protein > 1 g/dl and absence of: hollowed out areas of bone, Hypercalcemia (Calcium-serum < 11.5 mg/dl), Renal Failure (creatinine < 2 mg/dl) and anaemia (Hb > 10 g/dl or at least 2g/dl under normal value.
  * Alternatively, patients with Bone Marrow infiltration with CPs ≥ 10 %, or Ig G ≥ 3 g/dl or Ig A ≥ 2 g/dl or Bence Jones Protein > 1 g/24h (but not the two of them together) and always without: lytic lesions, Hypercalcaemia, Renal Failure and Anaemia could be admitted with the following additional criteria:

    * % CPs abnormal (CPa/CpcMO) ≥ 95 % with immunodeficiency, defined as diminution of levels of one or two Immunoglobulins of more than 25% respect normal values.
* ECOG >= 2.
* The patient has to be able to complain with the protocol visits.
* Women of childbearing age must have a negative pregnancy test during the 14 days before first dose. And they must accept to use anticonceptive methods beginning during all the study until 4 weeks after the last one.

Exclusion Criteria:

* Any other organic or mental illness that could make impossible to sign the Inform consent.
* Patients previously received treatment to smoldering Multiple Myeloma.
* Pregnancy or breast-feed women
* Hollowed out areas of bone, anaemia, renal failure and Hypercalcemia
* The following laboratory data:

  * Absolute neutrophil count ≥ 1000/mm3
  * Platelet count ≥ 75000/mm3
  * Aspartate transaminase (AST) or Alanine transaminase (ALT ) ≤ 3 x the upper limit of normal.
  * Total bilirubin: ≤ 2 x the upper limit of normal.
* Patients with >= Grade 2 peripheral neuropathy within 14 days before enrolment.
* Patient with a previous clinical history of another malignant illness except for squamous cell carcinoma or skin cancer or cervical cancer except the patient could be free of symptoms during ≥ 5 years.
* Patient has hypersensitivity or adverse events previous to lenalidomide or Dexamethasone.
* Patient who has major surgery during the 4th weeks previous inclusion.
* Patient has received other investigational drugs within 30 days before enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate when Revlimid and Dexamethasone treatment extend the time to progression to symptomatic MM in patients with smoldering MM | one year

SECONDARY OUTCOMES:
Evaluate the efficacy of the treatment in response rate terms | one year
Evaluate the safety and tolerability of the treatment | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mª Victoria Mateos, Dr, Principal Investigator — Hospital Clinico Universitario de Salamanca; Jesús San Miguel, Dr, Principal Investigator — Hospital Clínico Universitario de Salamanca; Joan Bladé, Dr, Principal Investigator — Hospital Clinic of Barcelona; Juan José Lahuerta, Dr, Principal Investigator — HOSPITAL DOCE DE OCTUBRE
Locations (13):
- Spain (13):
  - Hospital germans Trias i Pujol, Badalona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del SAS de Jerez de la Frontera, Jerez de la Frontera
  - Hospital de la Princesa, Madrid
  - Hospital Dode de Octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital General Univeristario Morales Messeguer, Murcia
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clínico de Valencia, Valencia
  - Hospital Universitario la Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] International Myeloma Working Group. Criteria for the classification of monoclonal gammopathies, multiple myeloma and related disorders: a report of the International Myeloma Working Group. Br J Haematol. 2003 Jun;121(5):749-57. PMID 12780789
- [Background] Dimopoulos MA, Moulopoulos A, Smith T, Delasalle KB, Alexanian R. Risk of disease progression in asymptomatic multiple myeloma. Am J Med. 1993 Jan;94(1):57-61. doi: 10.1016/0002-9343(93)90120-e. PMID 8420300
- [Background] Rajkumar SV. MGUS and smoldering multiple myeloma: update on pathogenesis, natural history, and management. Hematology Am Soc Hematol Educ Program. 2005:340-5. doi: 10.1182/asheducation-2005.1.340. PMID 16304401
- [Background] Wisloff F, Andersen P, Andersson TR, Brandt E, Eika C, Fjaestad K, Ly B, Lovasen K, Strom BR, Tjonnfjord GE. Has the incidence of multiple myeloma in old age been underestimated? The myeloma project of health region I in Norway. I. Eur J Haematol. 1991 Nov;47(5):333-7. doi: 10.1111/j.1600-0609.1991.tb01856.x. PMID 1761118
- [Background] Weber DM, Dimopoulos MA, Moulopoulos LA, Delasalle KB, Smith T, Alexanian R. Prognostic features of asymptomatic multiple myeloma. Br J Haematol. 1997 Jun;97(4):810-4. doi: 10.1046/j.1365-2141.1997.1122939.x. PMID 9217181
- [Background] Cesana C, Klersy C, Barbarano L, Nosari AM, Crugnola M, Pungolino E, Gargantini L, Granata S, Valentini M, Morra E. Prognostic factors for malignant transformation in monoclonal gammopathy of undetermined significance and smoldering multiple myeloma. J Clin Oncol. 2002 Mar 15;20(6):1625-34. doi: 10.1200/JCO.2002.20.6.1625. PMID 11896113
- [Background] Dimopoulos MA, Moulopoulos LA, Maniatis A, Alexanian R. Solitary plasmacytoma of bone and asymptomatic multiple myeloma. Blood. 2000 Sep 15;96(6):2037-44. PMID 10979944
- [Background] Rosinol L, Blade J, Esteve J, Aymerich M, Rozman M, Montoto S, Gine E, Nadal E, Filella X, Queralt R, Carrio A, Montserrat E. Smoldering multiple myeloma: natural history and recognition of an evolving type. Br J Haematol. 2003 Nov;123(4):631-6. doi: 10.1046/j.1365-2141.2003.04654.x. PMID 14616966
- [Background] Moulopoulos LA, Dimopoulos MA, Smith TL, Weber DM, Delasalle KB, Libshitz HI, Alexanian R. Prognostic significance of magnetic resonance imaging in patients with asymptomatic multiple myeloma. J Clin Oncol. 1995 Jan;13(1):251-6. doi: 10.1200/JCO.1995.13.1.251. PMID 7799027
- [Background] Perez-Persona E, Vidriales MB, Mateo G, Garcia-Sanz R, Mateos MV, de Coca AG, Galende J, Martin-Nunez G, Alonso JM, de Las Heras N, Hernandez JM, Martin A, Lopez-Berges C, Orfao A, San Miguel JF. New criteria to identify risk of progression in monoclonal gammopathy of uncertain significance and smoldering multiple myeloma based on multiparameter flow cytometry analysis of bone marrow plasma cells. Blood. 2007 Oct 1;110(7):2586-92. doi: 10.1182/blood-2007-05-088443. Epub 2007 Jun 18. PMID 17576818
- [Background] Hjorth M, Hellquist L, Holmberg E, Magnusson B, Rodjer S, Westin J. Initial versus deferred melphalan-prednisone therapy for asymptomatic multiple myeloma stage I--a randomized study. Myeloma Group of Western Sweden. Eur J Haematol. 1993 Feb;50(2):95-102. doi: 10.1111/j.1600-0609.1993.tb00148.x. PMID 8440364
- [Background] Rajkumar SV, Gertz MA, Lacy MQ, Dispenzieri A, Fonseca R, Geyer SM, Iturria N, Kumar S, Lust JA, Kyle RA, Greipp PR, Witzig TE. Thalidomide as initial therapy for early-stage myeloma. Leukemia. 2003 Apr;17(4):775-9. doi: 10.1038/sj.leu.2402866. PMID 12682636
- [Background] D'Amato RJ, Loughnan MS, Flynn E, Folkman J. Thalidomide is an inhibitor of angiogenesis. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):4082-5. doi: 10.1073/pnas.91.9.4082. PMID 7513432
- [Background] Geitz H, Handt S, Zwingenberger K. Thalidomide selectively modulates the density of cell surface molecules involved in the adhesion cascade. Immunopharmacology. 1996 Mar;31(2-3):213-21. doi: 10.1016/0162-3109(95)00050-x. PMID 8861747
- [Background] Haslett PA, Corral LG, Albert M, Kaplan G. Thalidomide costimulates primary human T lymphocytes, preferentially inducing proliferation, cytokine production, and cytotoxic responses in the CD8+ subset. J Exp Med. 1998 Jun 1;187(11):1885-92. doi: 10.1084/jem.187.11.1885. PMID 9607928
- [Background] Corral LG, Haslett PA, Muller GW, Chen R, Wong LM, Ocampo CJ, Patterson RT, Stirling DI, Kaplan G. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. J Immunol. 1999 Jul 1;163(1):380-6. PMID 10384139
- [Background] Parman T, Wiley MJ, Wells PG. Free radical-mediated oxidative DNA damage in the mechanism of thalidomide teratogenicity. Nat Med. 1999 May;5(5):582-5. doi: 10.1038/8466. PMID 10229238
- [Background] Davies FE, Raje N, Hideshima T, Lentzsch S, Young G, Tai YT, Lin B, Podar K, Gupta D, Chauhan D, Treon SP, Richardson PG, Schlossman RL, Morgan GJ, Muller GW, Stirling DI, Anderson KC. Thalidomide and immunomodulatory derivatives augment natural killer cell cytotoxicity in multiple myeloma. Blood. 2001 Jul 1;98(1):210-6. doi: 10.1182/blood.v98.1.210. PMID 11418482
- [Background] Richardson PG, Schlossman RL, Weller E, Hideshima T, Mitsiades C, Davies F, LeBlanc R, Catley LP, Doss D, Kelly K, McKenney M, Mechlowicz J, Freeman A, Deocampo R, Rich R, Ryoo JJ, Chauhan D, Balinski K, Zeldis J, Anderson KC. Immunomodulatory drug CC-5013 overcomes drug resistance and is well tolerated in patients with relapsed multiple myeloma. Blood. 2002 Nov 1;100(9):3063-7. doi: 10.1182/blood-2002-03-0996. PMID 12384400
- [Background] 20. Zangari M, Tricot G, Zeldis J, et al. Results of phase I study of CC-5013 for the treatment of multiple myeloma patients who relapse after high dose chemotherapy (HDCT). Blood 2001; 98:775a (Abstract 3226)
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] 23. Baz R, Choueiri TK, Jawde RA, et al. Doxil (D), Vincristine (V), Reduced Frequency Dexamethasone (d) and Revlimid(R) (DVd-R) Results in a High Response Rate in Patients with Refractory Multiple Myeloma(RMM).Blood 2005; 106: 2559.
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Hideshima T, Xiao H, Esseltine D, Schenkein D, Anderson KC; SUMMIT Investigators. Clinical factors predictive of outcome with bortezomib in patients with relapsed, refractory multiple myeloma. Blood. 2005 Nov 1;106(9):2977-81. doi: 10.1182/blood-2005-02-0691. Epub 2005 Jul 14. PMID 16020506
- [Background] Rajkumar SV, Hayman SR, Lacy MQ, Dispenzieri A, Geyer SM, Kabat B, Zeldenrust SR, Kumar S, Greipp PR, Fonseca R, Lust JA, Russell SJ, Kyle RA, Witzig TE, Gertz MA. Combination therapy with lenalidomide plus dexamethasone (Rev/Dex) for newly diagnosed myeloma. Blood. 2005 Dec 15;106(13):4050-3. doi: 10.1182/blood-2005-07-2817. Epub 2005 Aug 23. PMID 16118317
- [Background] Desikan R, Barlogie B, Sawyer J, Ayers D, Tricot G, Badros A, Zangari M, Munshi NC, Anaissie E, Spoon D, Siegel D, Jagannath S, Vesole D, Epstein J, Shaughnessy J, Fassas A, Lim S, Roberson P, Crowley J. Results of high-dose therapy for 1000 patients with multiple myeloma: durable complete remissions and superior survival in the absence of chromosome 13 abnormalities. Blood. 2000 Jun 15;95(12):4008-10. PMID 10845942
- [Background] 27. Palumbo A, Falco P, Musto P, et al. Oral RevlimidR Plus Melphalan and Prednisone (R-MP) for Newly Diagnosed Multiple Myeloma. Blood 2005; 106: 785.
- [Derived] Mateos MV, Hernandez MT, Salvador C, Rubia J, de Arriba F, Lopez-Corral L, Rosinol L, Paiva B, Palomera L, Bargay J, Oriol A, Prosper F, Lopez J, Arguinano JM, Blade J, Lahuerta JJ, San-Miguel J. Lenalidomide-dexamethasone versus observation in high-risk smoldering myeloma after 12 years of median follow-up time: A randomized, open-label study. Eur J Cancer. 2022 Oct;174:243-250. doi: 10.1016/j.ejca.2022.07.030. Epub 2022 Sep 5. PMID 36067617
- [Derived] Mateos MV, Hernandez MT, Giraldo P, de la Rubia J, de Arriba F, Corral LL, Rosinol L, Paiva B, Palomera L, Bargay J, Oriol A, Prosper F, Lopez J, Arguinano JM, Quintana N, Garcia JL, Blade J, Lahuerta JJ, Miguel JS. Lenalidomide plus dexamethasone versus observation in patients with high-risk smouldering multiple myeloma (QuiRedex): long-term follow-up of a randomised, controlled, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1127-1136. doi: 10.1016/S1470-2045(16)30124-3. Epub 2016 Jul 9. PMID 27402145
- [Derived] Paiva B, Mateos MV, Sanchez-Abarca LI, Puig N, Vidriales MB, Lopez-Corral L, Corchete LA, Hernandez MT, Bargay J, de Arriba F, de la Rubia J, Teruel AI, Giraldo P, Rosinol L, Prosper F, Oriol A, Hernandez J, Esteves G, Lahuerta JJ, Blade J, Perez-Simon JA, San Miguel JF; Spanish Myeloma Group / Program Study and Treatment of Hematological Malignancies cooperative study groups. Immune status of high-risk smoldering multiple myeloma patients and its therapeutic modulation under LenDex: a longitudinal analysis. Blood. 2016 Mar 3;127(9):1151-62. doi: 10.1182/blood-2015-10-662320. Epub 2015 Dec 14. PMID 26668134
- [Derived] Mateos MV, Hernandez MT, Giraldo P, de la Rubia J, de Arriba F, Lopez Corral L, Rosinol L, Paiva B, Palomera L, Bargay J, Oriol A, Prosper F, Lopez J, Olavarria E, Quintana N, Garcia JL, Blade J, Lahuerta JJ, San Miguel JF. Lenalidomide plus dexamethasone for high-risk smoldering multiple myeloma. N Engl J Med. 2013 Aug 1;369(5):438-47. doi: 10.1056/NEJMoa1300439. PMID 23902483
- [Derived] Matarraz S, Paiva B, Diez-Campelo M, Lopez-Corral L, Perez E, Mateos MV, Giraldo P, Hernandez MT, San Miguel JF, Orfao A; GEM Grupo Espanol de MM/Programa para el Estudio de la Terapeutica en Hemopatias Malignas Co-operative Study Groups. Myelodysplasia-associated immunophenotypic alterations of bone marrow cells in myeloma: are they present at diagnosis or are they induced by lenalidomide? Haematologica. 2012 Oct;97(10):1608-11. doi: 10.3324/haematol.2012.064121. Epub 2012 Apr 17. PMID 22511492
- [Derived] Weiss BM, Kuehl WM. Advances in understanding monoclonal gammopathy of undetermined significance as a precursor of multiple myeloma. Expert Rev Hematol. 2010 Apr;3(2):165-74. doi: 10.1586/ehm.10.13. PMID 20473362
- See also: Spanish association of Haematology — http://www.aehh.org